CLINICAL TRIAL: NCT03786822
Title: Reduction of Radiation Dose and Contrast Use During Cryoballoon Pulmonary Vein Isolation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Richard Wu, Professor of Internal Medicine, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 042013-074
Record Dates: First submitted 2018-11-29; First posted 2018-12-26 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Atrial Fibrillation
Keywords: cryoballoon; Atrial fibrillation; pulmonary vein isolation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Condition or Disease: Paroxysmal atrial fibrillation
  Procedure: Cryoballoon Pulmonary Vein Isolation
Who Masked: Outcomes Assessor
Masking Description: Subjects will be randomized in a 2:1 fashion
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non-fluoroscopic Cryoballoon PVI (Experimental): 1. Observation of pressure waveform change at the tip of the cryoballoon catheter from left atrial pressure to pulmonary vein pressure waveform.
  2. Intracardiac echocardiography (ICE) imaging with no Doppler color evidence of peri-balloon high velocity leaks.
  3. Intracardiac echo imaging showing no evidence of leak during agitated saline contrast injection into cryoballoon catheter positioned at pulmonary vein ostium.
  Interventions: Procedure: Cryoballoon Pulmonary Vein Isolation - PVI
- Fluoroscopic Cryoballoon PVI (Active Comparator): Standard cryoballoon PVI using radio opaque contrast pulmonary vein angiography
  Interventions: Procedure: Cryoballoon Pulmonary Vein Isolation - PVI

INTERVENTIONS:
Procedure: Cryoballoon Pulmonary Vein Isolation - PVI — A 28-mm cryoballoon (Arctic Front Advance™ Cardiac CryoAblation Catheter, Medtronic, Minneapolis, MN) will be employed. The cryoballoon catheter will be introduced into the left atrium, following a single transeptal puncture, through a 12 French steerable sheath (FlexCath, Medtronic), constantly flushed with heparinized saline. A circular mapping catheter (Achieve, Medtronic) will be advanced through the cryoballoon to the PV orifice and positioned as proximally as possible inside the vessel to record the PV potentials at baseline and monitor the isolation procedure in real time.
  Other Names: Atrial Fibrillation Ablation

SUMMARY:
This is a multi-site, randomized, investigator-initiated pilot study to evaluate the efficacy of investigational techniques to reduce fluoroscopy time or radiation dose and the amount of radio opaque contrast used during a cryoballoon pulmonary vein isolation procedure for atrial fibrillation.

One group of subjects will have the procedure performed with intracardiac echo maneuvers to assess cryoballoon occlusion of the pulmonary vein and will be compared to a group of subjects who will receive the standard medical treatment with fluoroscopy and angiography.

DETAILED DESCRIPTION:
Surgical and catheter based technologies target triggers that initiate atrial fibrillation located in the pulmonary veins (PV). In order to isolate these triggers, radiofrequency energy or freezing is used to destroy the atrial tissue which propagate electrical impulses into and out of the pulmonary veins (PV), to achieve pulmonary vein isolation (PVI). Use of a patented cryoballoon catheter (Medtronic) to perform PVI has been shown to be safe and efficacious under fluoroscopic guidance with contrast angiography. The objective of this study is to identify methods to reduce radiation dose and radio opaque contrast use while maintaining PVI efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal atrial fibrillation refractory to treatment with anti-arrhythmic drugs
* Must be able to undergo pre-operative cardiac CT angiogram or cardiac MRI to define pulmonary vein anatomy.

Exclusion criteria:

* Planned use of radiofrequency cardiac ablation
* Presence of a cardiac implantable electronic device
* Conditions where manipulation of the catheter would be unsafe such as intracardiac thrombus
* Patients with active systemic infections
* Patients with cryoglobulinemia
* Pregnant and/or breast-feeding females are excluded from this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Reduction of Radiation Dose during Cryoballoon Pulmonary Vein Isolation. | one year
  change in the composite endpoint of total fluoroscopy time (min)
Reduction of Contrast during Cryoballoon Pulmonary Vein Isolation. | one year
  change in the composite endpoint of contrast (cc)

SECONDARY OUTCOMES:
Recurrence of atrial fibrillation | one year
  •recurrence of atrial fibrillation after 1 month blanking period measured by ECG event monitoring at 6 and 12 month follow up (time to first recurrence in months, total number of episodes, and total duration in hours)
Time to Cryoballoon Pulmonary Vein Isolation | one year
  •cryoballoon procedure time (min)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States